CLINICAL TRIAL: NCT01713634
Title: Dietary Intake Can Predict and Protect Against Changes in Bone Metabolism During Spaceflight and Recovery
Brief Title: Dietary Intake Modifications to Protect Against Changes in Bone Metabolism
Acronym: ProK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Scott M. Smith, Manager for Nutritional Biochemistry, National Aeronautics and Space Administration (NASA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Pro0225
Record Dates: First submitted 2012-10-19; First posted 2012-10-25 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Bone Resorption
Keywords: Bone resorption; Diet
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Apro/K Diet (Experimental): Subjects consume a prescribed diet for 4 days with a low ratio of animal protein to potassium (0.3-0.6 g/mEq).
  Interventions: Other: Preflight; Other: In-flight
- High Apro/K Diet (Experimental): Subjects consume a prescribed diet that has a high ratio of animal protein to potassium (1.0-1.3 g/mEq) for 4 days.
  Interventions: Other: Preflight; Other: In-flight

INTERVENTIONS:
Other: Preflight — 4-d controlled diet sessions will occur twice before flight.
Other: In-flight — 4-d controlled diet sessions will take place on flight days 15, 60, 120, and 180. Flight day 30 will only be monitored intakes (subject consume nominal intake)

SUMMARY:
Bone loss is not only a well-documented effect of spaceflight on astronauts, but also a condition that affects millions of men and women on Earth each year. Many countermeasures to bone loss have been proposed, and many have been evaluated to some degree. To date, those showing potential have focused on either exercise or pharmacological interventions, but none have targeted dietary intake alone as a factor to predict or minimize bone loss during spaceflight. The investigators proposed to document how the ratio of acid precursors to base precursors in the diet is related to directional changes in markers of bone resorption and formation during flight and recovery from flight. There is a high likelihood for success in predicting the extent of bone loss from dietary intake patterns of astronauts during spaceflight, given that this concept is strongly anchored in data obtained from ground-based experiments in our laboratory and others. The notion of manipulating diet to minimize bone loss could also have significant social and economic impacts for NASA and for the general public - especially given the increasing trends for diets that are high in animal protein and low in fruits and vegetables. The results of the proposed experiments will lead to development of a dietary countermeasure for bone loss consisting of a balanced diet with no associated risks for side effects that might be present with pharmaceuticals or supplements, no requirement for payload mass, and no additional crew time necessary during flight.

ELIGIBILITY:
Inclusion Criteria:

* Astronauts flying on long-duration (3-6 months) spaceflights

Exclusion Criteria:

* Non-astronauts

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in urinary n-telopeptide after 15 days of space flight compared to preflight | 15 days
  24-h NTX will be used as an indicator of bone resorption
Change in urinary n-telopeptide after 30 days of space flight compared to preflight | 30 days
Change in urinary n-telopeptide after 60 days of space flight compared to preflight | 60 days
Change in urinary n-telopeptide after 120 days of space flight compared to preflight | 120 days
Change in urinary n-telopeptide after 180 days of space flight compared to preflight | 180 days
Change in urinary calcium after 15 days of space flight compared to preflight | 15 days
Change in urinary calcium after 60 days of space flight compared to preflight | 60 days
Change in urinary calcium after 120 days of space flight compared to preflight | 120 days
Change in urinary calcium after 180 days of space flight compared to preflight | 180 days

SECONDARY OUTCOMES:
Change in urinary calcium after 30 days of space flight compared to preflight | 30 days
  24-h urinary calcium

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Smith, PhD, Principal Investigator — National Aeronautics and Space Administration (NASA)
Locations (1):
- Johnson Space Center, Houston, Texas, United States

REFERENCES:
- [Background] Zwart SR, Hargens AR, Smith SM. The ratio of animal protein intake to potassium intake is a predictor of bone resorption in space flight analogues and in ambulatory subjects. Am J Clin Nutr. 2004 Oct;80(4):1058-65. doi: 10.1093/ajcn/80.4.1058. PMID 15447920
- [Background] Zwart SR, Davis-Street JE, Paddon-Jones D, Ferrando AA, Wolfe RR, Smith SM. Amino acid supplementation alters bone metabolism during simulated weightlessness. J Appl Physiol (1985). 2005 Jul;99(1):134-40. doi: 10.1152/japplphysiol.01406.2004. Epub 2005 Feb 3. PMID 15691900
- [Derived] Zwart SR, Rice BL, Dlouhy H, Shackelford LC, Heer M, Koslovsky MD, Smith SM. Dietary acid load and bone turnover during long-duration spaceflight and bed rest. Am J Clin Nutr. 2018 May 1;107(5):834-844. doi: 10.1093/ajcn/nqy029. PMID 29722847